CLINICAL TRIAL: NCT04109352
Title: Validation and Field-applicability of a 13C-Sucrose Breath Test to Assess Carbohydrate Uptake and Utilization in Environmental Enteropathy Among Children in Resource Poor Settings: A Multi-site Prospective Study
Brief Title: Labelled Carbon Sucrose Breath Test (13C-SBT) as a Marker of Environmental Enteropathy
Acronym: SBT4EE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Collaborators: International Atomic Energy Agency (Other Government); Flinders University (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); St. John's Research Institute (Other); The University of The West Indies (Other); Mmust Masinde Muliro University of Science and Technology (Unknown); Asociacion Benefica Prisma (Other); Scottish Universities Environmental Research Centre (Other); University of Michigan (Other); Tropical Diseases Research Centre, Zambia (Other Government); Gastroenterology Services, Ltd. (Other)
Responsible Party: Principal Investigator, Margaret Kosek, MD, Associate Professor, University of Virginia
Other Study IDs: CE0783.19
Record Dates: First submitted 2019-07-20; First posted 2019-09-30 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Glucose-Galactose Malabsorption; Enteropathy; Malnutrition, Child; Intestinal Permeability; Linear Growth Failure
MeSH Terms: conditions — Glucose-Galactose Malabsorption; Intestinal Diseases; Child Nutrition Disorders; Failure to Thrive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breath prior to and following enriched sucrose ingestion, plasma, saliva, stool, urine following the ingestion of rhamnose and lactulose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Linear growth failure, a manifestation of chronic undernutrition in early childhood, is a recalcitrant problem in resource constrained settings. The underlying causes of growth failure are multifactorial, but persistent and recurrent infection and inflammation of the gastrointestinal tract and immune activation, a condition commonly referred to as environmental enteropathy, is an important contributor. A highly enriched 13C-Sucrose Breath Test, a measure of sucrase-isomaltase activity, will be evaluated as a non-invasive biomarker of environmental enteropathy, and more specifically of intestinal brush border enzyme activity in 6 resource poor countries (Bangladesh, India, Jamaica, Kenya, Peru and Zambia) in 100 volunteers aged 12-15 months (total n=600) and evaluated relative to the lactose rhamnose test and linear and ponderal growth over a 3-6 month period following biomarker assessment. Field usability will also be assessed.

DETAILED DESCRIPTION:
Environmental enteropathy is associated with linear and ponderal growth shortfalls in young children in resource constrained settings. However, the physiological alterations of intestinal function that accompany both the demonstrable evidence of inflammation and architectural changes seen in biopsies from effected children have yet to be elucidated, and this knowledge gap limits the development of effective strategies to optimally manage the condition. Furthermore, a limited number of non-invasive assays exist with which to assess the presence of environmental enteropathy in low resource settings. This study aims 1) to determine if sucrose-isomaltase enzyme is altered in children with environmental enteropathy by using a 13C-Sucrose breath test 2) to determine if the test is able to be employed in resource limited settings.

ELIGIBILITY:
Inclusion Criteria:

All children will be recruited and enrolled through convenience sampling, either at the community level (if the study site has previously censused the community) or through child clinic visits.

Exclusion Criteria:

1. Severe acute malnutrition
2. HIV positive
3. Weight for height Z >+2
4. Known medical illness contributing to growth failure

Ages: 12 Months to 15 Months | Sex: All
Age Groups: Child
Study Population: Because of exigent test requirements enrollment will be restricted to convenience samples from populations near centers of excellence in nutritional studies in Dhaka, Bangladesh (the International Centre for Diarrhoeal Disease Research); Bangalore, India (St. John's Research Institute, St. John's National Academy of Health Sciences); Kingston, Jamaica (The Tropical Metabolism Research Unit of the Caribbean Institute for Health Research, University of West Indies); Kakamega, Kenya (Masinde Muliro University of Science and Technology); Iquitos, Peru44 (Asociación Benefica PRISMA and the University of Virginia); and Ndola, Zambia (Tropical Disease Research Centre). These sites represent a range of epidemiologic contexts which will enhance the cross-context applicability of study results.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of SBT to Lactulose rhamnose (LR) test-% dose 90 min | 6 months after enrollment is completed
  The 13C-SBT (cumulative percent of dose recovered at 90 minutes post administration) will be compared to LR ratio (the ratio of the percent recovery of administered lactulose and mannitol)
Comparison of SBT to Lactulose rhamnose (LR) test- time to 50% recovery | 6 months after enrollment is completed
  The 13C-SBT (time to 50% area under the curve of 13C tracer, expressed in minutes ) will be compared to LR ratio (the ratio of the percent recovery of administered lactulose and mannitol)
Correlation of SBT (% recovery at 90 minutes) to Lactulose rhamnose (LR) test-Lactulose recovery | 6 months after enrollment is completed
  The 13C-SBT (cumulative percent of dose recovered at 90 minutes post administration) will be compared to the percent lactulose recovery at 90 minutes post administration
Correlation of SBT (time to 50% recovery) to Lactulose rhamnose (LR) test-Lactulose recovery | 6 months after enrollment is completed
  The 13C-SBT (time to 50% area under the curve 13C tracer, expressed in minutes) will be compared to the percent lactulose recovery at 90 minutes post administration
Correlation of SBT (% dose recovered at 09 minutes) to Lactulose rhamnose (LR) test-Mannitol recovery | 6 months after enrollment is completed
  The 13C-SBT (cumulative percent of dose of 13C recovered at 90 minutes post administration) will be compared to percent mannitol recovery
Correlation of SBT (time to recovery of 50% of dose) to Lactulose rhamnose (LR) test-Mannitol recovery | 6 months after enrollment is completed
  The 13C-SBT (time to 50% area under the curve 13C tracer, expressed in minutes) will be compared to percent mannitol recovery
Characterize the relationship between SBT (% of dose recovered at 90 min) and baseline childhood anthropometrics (attained length) | 6 months after enrollment is completed
  We will compare results of the SBT test expressed as cumulative percent of dose recovered at 90 minutes post administration and LAZ (length for age Z-score as defined by 2006 World Health Organization norms, cross-sectional)
Characterize the relationship between SBT (time to recovery of 50% of dose) and baseline childhood anthropometrics (attained length) | 6 months after enrollment is completed
  We will compare results of the SBT test expressed as time to 50% area under the curve 13C tracer, expressed in minutes and LAZ (length for age Z-score as defined by 2006 World Health Organization norms, cross-sectional)
Characterize the relationship between SBT and childhood anthropometrics (attained weight) | 6 months after enrollment is completed
  We will compare results of the SBT test expressed as the cumulative percent of dose recovered at 90 minutes post administration and WAZ (weight for age Z-score as defined by 2006 World Health Organization norms, cross-sectional)
Characterize the relationship between SBT and childhood anthropometrics (attained weight for height) | 6 months after enrollment is completed
  We will compare results of the SBT test expressed as time to 50% area under the curve 13C tracer, expressed in minutes and WAZ (weight for age Z-score as defined by 2006 World Health Organization norms, cross-sectional)
Characterize the relationship between SBT (time to 50% recovery of 13C) and childhood linear growth, 3 months | 6 months after enrollment is completed
  We will compare values for the 13C-SBT expressed as time to 50% area under the curve 13C tracer, expressed in minutes and change in length for age Z score (WHO 2006 reference standards) over the subsequent 3 months
Characterize the relationship between SBT and childhood linear growth, 6 months | 6 months after enrollment is completed
  We will compare values for the 13C-SBT expressed as time to 50% area under the curve 13C tracer, expressed in minutes and change in length for age Z score (WHO 2006 reference standards) over the subsequent 6 months
Characterize the relationship between SBT (% dose recovered at 90 min)and childhood linear growth, 3 months | 6 months after enrollment is completed
  We will compare the 13C-SBT tests results (cumulative percent of dose recovered at 90 minutes post administration) and change in LAZ over the subsequent 3 months
Characterize the relationship between SBT and childhood linear growth | 6 months after enrollment is completed
  We will compare the 13C-SBT tests results (cumulative percent of dose recovered at 90 minutes post administration) and change in LAZ over the subsequent 6 months

SECONDARY OUTCOMES:
Assess the relationship between the 13C-SBT (% recovery 90min) and fecal myeloperoxidase | Six months from the enrollment of the last subject
  Compare fecal myeloperoxidase concentration (ng/mL) with 13SBT (% of cumulative dose recovered at 90 minutes, expressed as %)
Assess the relationship between SBT ( time to recovery of 50% of the 13C-tracer) and fecal myeloperoxidase | Six months from the enrollment of the last subject
  Compare fecal myeloperoxidase concentration (ng/mL) with 13SBT (time to recovery of 50% of the administered 13C tracer, measured in minutes)
Assess the relationship between the 13C-SBT (% recovery 90 min) and serum fatty acid binding protein | Six months from the enrollment of the last subject
  Compare serum fatty acid binding protein concentration (ng/mL), with 13SBT as assessed by % of administered dose recovered at 90 minutes
Assess the relationship between the 13C-SBT (time to 50% recovery) and serum fatty acid binding protein concentration | Six months from the enrollment of the last subject
  Compare serum fatty acid binding protein concentration (ng/mL) with 13SBT as measured by the time (in minutes) to the recovery of 50% of the administered dose of 13C.
Assess the relationship between the 13C-SBT (time to 50% recovery) and kynurenine tryptophan ratio | Six months from the enrollment of the last subject
  Compare time to recovery of 50% of 13C probe of SBT with kynurenine tryptophan ratio (molar ratio of KT multiplied by 1000)
Assess the relationship between the 13C-SBT (% recovery at 90 minutes) and kynurenine tryptophan ratio, | Six months from the enrollment of the last subject
  Compare 13C SBT as measured by % recovery of 13C probe at 90 minutes with kynurenine tryptophan ratio
Assess the relationship between the 13C-SBT as assessed by percent of 13C tracer recovered in at 90 minutes and fecal alpha-antitrypsin concentration | Six months from the enrollment of the last subject
  Compare 13CSBT as measured by the percent of tracer recovered at 90 minutes with fecal anti-trypsin concentration (mg/g)
Assess the relationship between the 13C-SBT as measured by the time to 50% recovery of 13C and fecal alpha-antitrypsin | Six months from the enrollment of the last subject
  Compare 13C SBT as measured by the time to 50% recovery of 13C with fecal anti-trypsin concentration (mg/g)

OTHER OUTCOMES:
Reproducibility of the 13C-SBT test , percent of dose recovered in first 90 minutes | Six months from the enrollment of the last subject
  We will assess the coefficient of variation and correlation coefficient between repeated cumulative percent of dose recovered at 90 minutes post administration on separate SBT tests administered one week apart done on the same child (Peru site only).
Reproducibility of the 13C-SBT test, time to 50% area under the curve of 13C tracer, expressed in minutes | Six months from the enrollment of the last subject
  We will assess the coefficient of variation and correlation coefficient between repeated SBT tests 7 days apart as assessed by the time to 50% area under the curve of 13C tracer, expressed in minutes from the same child (Peru site only).
Epidemiologic factors that influence 13C-SBT measure, percent of dose recovered at 90 minutes | Six months from the enrollment of the last subject
  Determine if significant associations exist between 13C-SBT measured as cumulative percent of dose recovered at 90 minutes post administration and the WAMI index.The WAMI index is a previously validated composite index of environmental variables to create a index that expresses the socioeconomic and physical environment in diverse geographical contexts (PMID 24656134)
Epidemiologic factors that influence 13C-SBT measure, time to 50% AUC recovered | Six months from the enrollment of the last subject
  Determine if significant associations exist between 13C-SBT measured as the time to recovery of 50% of the administered tracer and the WAMI index. The WAMI index is a previously validated composite index of environmental variables to create a index that expresses the socioeconomic and physical environment in diverse geographical contexts ((PMID 24656134).

CONTACTS AND LOCATIONS:
Overall Officials: Victor Owino, PhD, Study Chair — International Atomic Energy Agency
Locations (9):
- Flinders University, Adelaide, Australia
- Nutrition and Clincial Services Division, icddr, b, Dhaka, Bangladesh
- CBCI Society for Medical Education, St John's Research Institute, Bengaluru, India
- Tropical Metabolism Research Unit, University of West Indies, Kingston, Jamaica
- Masinde Muliro University of Science and Technology, Kakamega, Kenya
- Investigaciones Biomedicas, Asociacion Benefica PRISMA, Iquitos, Peru
- Scottish Universities Environmental Research Centre, East Kilbride, United Kingdom
- Zambia (2):
  - Tropical Gastroenterology & Nutrition Ltd, Lusaka
  - Tropical Diseases Research Centre, Ndola

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shivakumar N, Huq S, Paredes-Olortegui M, Konyole SO, Devi S, Yazbeck R, Owino VO, Brouwer AF, Kosek MN, Kelly P, Morrison DJ, Lee GO. A cross-sectional study of associations between the 13C-sucrose breath test, the lactulose rhamnose assay, and growth in children at high risk of environmental enteropathy. Am J Clin Nutr. 2024 Dec;120(6):1354-1363. doi: 10.1016/j.ajcnut.2024.10.001. Epub 2024 Oct 9. PMID 39384142
- [Derived] Lee GO, Schillinger R, Shivakumar N, Whyte S, Huq S, Ochieng Konyole S, Chileshe J, Paredes-Olortegui M, Owino V, Yazbeck R, Kosek MN, Kelly P, Morrison D. Optimisation, validation and field applicability of a 13C-sucrose breath test to assess intestinal function in environmental enteropathy among children in resource poor settings: study protocol for a prospective study in Bangladesh, India, Kenya, Jamaica, Peru and Zambia. BMJ Open. 2020 Nov 17;10(11):e035841. doi: 10.1136/bmjopen-2019-035841. PMID 33203623